CLINICAL TRIAL: NCT04926051
Title: A Phase 1, Double-blind, Placebo-controlled, Randomized, Single and Multiple Ascending Dose, and a Japanese Multiple Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BMS-986172, Including an Open-Label Assessment of Relative Bioavailability and Food Effect on the Single-Dose Pharmacokinetics of BMS-986172 in Healthy and Obese Otherwise Healthy Participants
Brief Title: A Study to Assess the Safety, Tolerability and Drug Levels of BMS-986172 in Healthy and Obese Participants, Including an Assessment of the Effects of Food on BMS-986172 Absorption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MB008-009
Record Dates: First submitted 2021-06-11; First posted 2021-06-14 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; BMS-986172

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: SAD (Experimental): SAD = Single Ascending Dose
  Interventions: Drug: BMS-986172; Other: Placebo
- Part B: MAD (Experimental): MAD = Multiple Ascending Dose
  Interventions: Drug: BMS-986172; Other: Placebo
- Part C: JMAD (Experimental): JMAD= Japanese Multiple Ascending Dose
  Interventions: Drug: BMS-986172; Other: Placebo
- Part D: FE/BA (Experimental): FE/BA = Food Effect/Relative Bioavailability
  Interventions: Drug: BMS-986172

INTERVENTIONS:
Drug: BMS-986172 — Specified dose on specified days
Other: Placebo — Specified dose on specified days
  Arms: Part A: SAD; Part B: MAD; Part C: JMAD

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and drug levels of BMS-986172 and evaluate the effects of food on BMS-986172 absorption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as determined by no clinically significant deviation from normal in medical history, physical examination, vital signs, ECG, and clinical laboratory results as determined by the investigator or designee.
* Participants in Part C must be first-generation Japanese participants. For the purpose of this study, first-generation Japanese is defined as native Japanese or first-generation Japanese living outside of Japan for <10 years.
* BMI of ≥ 18 kg/m2 to ≤ 40.0 kg/m2, inclusive, at screening, except for high BMI cohort participants (Part B) which will be restricted to a BMI range of ≥ 30 kg/m2 to ≤ 40.0 kg/m2.

Exclusion Criteria:

* Inability to tolerate the oral lipid meal or the testing conditions on Day -1, including but not limited to: bloating, nausea, vomiting, diarrhea, pain, or any discomfort due to oral lipid meal.
* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or that may compromise the objectives of the study, including active, or history of, liver disease, or intestinal disorder including irritable bowel syndrome.
* History or presence of malignancy including hematological malignancies; participants with a history of basal cell or squamous cell carcinoma that has been treated with no evidence of recurrence within 5 years will be allowed for inclusion, as judged by the investigator or designee.
* Any significant acute or chronic medical illness.
* History of SARS-CoV-2 infection (either suspected or confirmed) within 3 months prior to signing consent
* Participants who have received a SARS-CoV-2 vaccine approved for Emergency Use Authorization by the US FDA that is not live attenuated may be considered for enrollment

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Incidence of non-serious Adverse Events (AEs) | Up to 35 days
Incidence of Serious Adverse Events (SAEs) | Up to 35 days
Incidence of AEs leading to discontinuation of study treatment | Up to 35 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 28 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 28 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 28 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 28 days
Incidence of clinically significant changes in physical examination | Up to 28 days
Incidence of clinically significant changes in clinical laboratory values: Hematology tests | Up to 28 days
Incidence of clinically significant changes in clinical laboratory values: Chemistry tests | Up to 28 days
Incidence of clinically significant changes in clinical laboratory values: Urinalysis tests | Up to 28 days
Incidence of clinically significant changes in clinical laboratory values: Serology tests | Up to 28 days
Incidence of clinically significant changes in ECG parameters: QTcF | Up to 28 days
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave

SECONDARY OUTCOMES:
Plasma concentrations of BMS-986172 | Up to 28 days
Maximum observed plasma concentration (Cmax) | Up to 28 days
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON Plc (Legacy PRA), Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm